CLINICAL TRIAL: NCT06634381
Title: Patient Descriptors Of Cancer-Related Fatigue: A Mixed Methods Pilot Study Of Cancer Survivors
Acronym: VAP
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00119101; ONC-CCS-2402 (Other: Atrium Health)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Fatigue
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Cancer survivors with any type of cancer and a history of at least 1 visit for the purpose of monitoring long term care post curative treatment at LCH and/or the Charlotte or Winston-Salem campuses of AHWFBCCC who have completed curative treatment for more than 6 months.
  Interventions: Behavioral: CRF Visual Aid
- Clinicians: Any providers working with post-treatment oncology survivors at LCH and the Charlotte or Winston Salem campuses of AHWFBCCC.
  Interventions: Behavioral: CRF Visual Aid

INTERVENTIONS:
Behavioral: CRF Visual Aid — After all qualitative interviews and associated quantitative data analysis are complete, the visual aid will be created to illustrate, through a type of Venn Diagram, how the data are related.

SUMMARY:
The purpose of this research study is to better understand how cancer-related fatigue affects patients and how it's discussed with providers. This information will be used to develop an educational resource (visual aid poster) that could help individuals and their providers talk about cancer-related fatigue and which may help individuals better manage this symptom.

DETAILED DESCRIPTION:
This is a mixed methods cross-sectional pilot study. The target population is adults ≥ 18 years of age who have been diagnosed with cancer, have completed anti-cancer treatment more than six months ago, have no current detectable evidence of cancer, and are experiencing cancer-related fatigue. Participation in this research will involve completion of a six-minute walk test, survey completion, two virtual video interviews, and potentially one additional virtual interview. The interviews will include two 45 minutes for survivors and one 30-minute interview for clinicians. An additional 30-minute interview will be conducted for each survivor and clinician group.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with study procedures for the duration of the study

Survivors:

* Written informed consent and HIPAA authorization for release of personal information
* Ability to read/write, understand and converse in English without the need for an interpreter
* Men and women aged ≥ 18 years at the time of consent
* White or Caucasian, Black or African American, or Hispanic or Latino/a
* History of at least one visit for the purpose of monitoring long term care post curative treatment at LCH and/or the Charlotte or Winston-Salem campuses of AHWFBCCC
* Completed curative treatment > 6 months ago for any cancer type, with no detectable evidence of cancer
* Self-reported fatigue score of ≥ 4 on the Numerical Rating Scale

Clinicians:

- Currently see oncology patients (any cancer type) for survivorship care at LCH and/or the Charlotte or Winston-Salem campuses of AHWFBCCC

Exclusion Criteria:

Survivors:

* Continuing maintenance therapy or other cancer-related treatment (i.e. immunotherapy or hormonal therapy)
* History of or current severe or untreated depression
* Hemoglobin <11g/dL at last CBC SOC lab collection
* History/diagnosis of dementia
* Factors or conditions, for which participation may (1) not be in the best interest or (2) interfere with study assessment results (e.g. medical comorbidities, primary brain tumor/metastases)
* No access to internet/Wi-Fi

Clinicians:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer survivors and clinicians at LCH and/or at the Charlotte or Winston-Salem campuses of AHWFBCCC.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Domains reflecting cancer-related fatigue (CRF) experiences in cancer survivors | Seven months from baseline
  A domain is a topic that people talk about that has sub-items characterizing the distinct features and levels of importance within the domain. Using qualitative analysis, evaluation of how survivors think and talk about CRF to generate domain classifications of language. Domain is a categorical variable.

SECONDARY OUTCOMES:
Qualitative themes derived from open-ended interviews of clinicians | Five months from screening
  Qualitative themes resulting from the inductive analysis of open-ended questions administered in clinician interviews. A qualitative theme is the outcome of coding, a label that reflects what a unit of data is about or what it means. Qualitative theme is categorical variable.
Domains reflecting CRF experiences in cancer survivors | Seven months from baseline
  Each domain is a binary variable to indicate whether the domain was used or not used.
Appropriateness of the visual aid to alleviate survivor-clinician communication barriers | Eleven months from baseline
  Appropriateness is the degree to which the visual aid addresses patients' needs for communicating CRF and clinicians' needs for assessing CRF. Appropriateness is an ordinal variable.

CONTACTS AND LOCATIONS:
Overall Officials: Dori Beeler, PhD, Principal Investigator — Atrium Health Wake Forest Baptist Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Levine Childrens Hospital Pediatric Cancer and Blood Disorders, Charlotte, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No